CLINICAL TRIAL: NCT03437538
Title: Reduction Ratio and Clearance of Middle Molecules During a Single Hemodialysis Session With Medium Cut-Off (MCO) Filter Compared to Hemodiafiltration (HDF) With Standard High-flux Filter
Brief Title: Reduction Ratio and Clearance During Hemodialysis With MCO-filter Compared to HDF With Standard High-flux Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017/830/1
Record Dates: First submitted 2018-01-22; First posted 2018-02-19 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Chronic Kidney Failure; Uremia; Dialysis
Keywords: Dialysis; MCO; Middle molecules; High Retention Onset; Medium Cut-Off
MeSH Terms: conditions — Kidney Failure, Chronic; Uremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First MCO-HD, then High-flux-HDF (Active Comparator): Participants with ongoing HDF-treatments will have measurements during an intervention with a 4h dialysis with MCO-HD, followed by 2 weeks of washout with ordinary HDF, thereafter measurements during a 4h dialysis with High-flux-HDF
  Interventions: Device: MCO-HD; Device: High-flux HDF
- First High-flux-HDF, then MCO-HD (Active Comparator): Participants with ongoing HDF-treatments will have measurements during a 4h dialysis with High-flux-HDF, followed by 2 weeks of washout with ordinary HDF, thereafter measurements during an intervention with a 4h dialysis with MCO-HD
  Interventions: Device: MCO-HD; Device: High-flux HDF

INTERVENTIONS:
Device: MCO-HD — Measurements will be done during a single hemodialysis session with Medium Cut-Off filter
Device: High-flux HDF — Measurements will be done during a single hemodiafiltration session with standard high-flux filter

SUMMARY:
The Medium Cut-Off dialysis (MCO) membrane has been developed to improve middle molecule removal compared to standard high-flux dialysis filters.

The major aim of this study is to compare the reduction ratio of middle molecules, during a single hemodialysis session with MCO-filter, compared to hemodiafiltration (HDF) with standard high-flux filter.

Secondary aims are to compare the reduction ratio of small and large molecules between the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing HDF treatment
* CRP <30
* No Acute Myocardial Infarction within 3 months.

Exclusion Criteria:

* Not able to understand the study information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Reduction ratio (RR) of middle molecules (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin) | 4 hours
  Reduction ratio during a 4h dialysis session. (Predialysis concentration - Postdialysis concentration)/Predialysis concentration*100%
Instantaneous arteriovenous clearance of middle molecules (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin) | 30 minutes
  Instantaneous arteriovenous clearance (ml/min) at 30 minutes of dialysis.
Instantaneous arteriovenous clearance of middle molecules (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin) | 60 minutes
  Instantaneous arteriovenous clearance (ml/min) at 60 minutes of dialysis.
Instantaneous arteriovenous clearance of middle molecules (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin) | 120 minutes
  Instantaneous arteriovenous clearance (ml/min) at 120 minutes of dialysis.
Instantaneous arteriovenous clearance of middle molecules (Beta-2-microglobulin, Cystatin C, Myoglobin, Beta-Trace Protein, Troponin T, Prealbumin) | 240 minutes
  Instantaneous arteriovenous clearance (ml/min) at 240 minutes of dialysis.

SECONDARY OUTCOMES:
RR of large molecules (Albumin, Transferrin, IgG) | 4 hours
  Reduction ratio during a 4h dialysis session. (Predialysis concentration - Postdialysis concentration)/Predialysis concentration*100%
RR of small molecules (Urea, Phosphate, Creatinine) | 4 hours
  Reduction ratio during a 4h dialysis session. (Predialysis concentration - Postdialysis concentration)/Predialysis concentration*100%
Number of Adverse Events | 4 hours
  Number of adverse events during a 4h dialysis session
Instantaneous arteriovenous clearance of large molecules (Albumin, Transferrin, IgG) | 30 minutes
  Instantaneous arteriovenous clearance (ml/min) at 30 minutes of dialysis.
Instantaneous arteriovenous clearance of large molecules (Albumin, Transferrin, IgG) | 60 minutes
  Instantaneous arteriovenous clearance (ml/min) at 60 minutes of dialysis.
Instantaneous arteriovenous clearance of large molecules (Albumin, Transferrin, IgG) | 120 minutes
  Instantaneous arteriovenous clearance (ml/min) at 120 minutes of dialysis.
Instantaneous arteriovenous clearance of large molecules (Albumin, Transferrin, IgG) | 240 minutes
  Instantaneous arteriovenous clearance (ml/min) at 240 minutes of dialysis.
Instantaneous arteriovenous clearance of small molecules (Urea, Phosphate, Creatinine) | 30 minutes
  Instantaneous arteriovenous clearance (ml/min) at 30 minutes of dialysis.
Instantaneous arteriovenous clearance of small molecules (Urea, Phosphate, Creatinine) | 60 minutes
  Instantaneous arteriovenous clearance (ml/min) at 60 minutes of dialysis.
Instantaneous arteriovenous clearance of small molecules (Urea, Phosphate, Creatinine) | 120 minutes
  Instantaneous arteriovenous clearance (ml/min) at 120 minutes of dialysis.
Instantaneous arteriovenous clearance of small molecules (Urea, Phosphate, Creatinine) | 240 minutes
  Instantaneous arteriovenous clearance (ml/min) at 240 minutes of dialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Christensson, MD, PhD, Principal Investigator — Region Skane, Lund University
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No